CLINICAL TRIAL: NCT03815110
Title: Preeclampsia Risk Assessment: Evaluation of Cut-offs to Improve Stratification
Acronym: PRAECIS
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: ThermoFisher Scientific Brahms Biomarkers France (Industry)
Responsible Party: Principal Investigator, S Ananth Karumanchi, Lead Principal Investigator, Cedars-Sinai Medical Center
Other Study IDs: Pro00055135
Record Dates: First submitted 2019-01-17; First posted 2019-01-24 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Preeclampsia and Eclampsia; Preeclampsia Severe; Gestational Hypertension; Chronic Hypertension in Obstetric Context; Superimposed Pre-Eclampsia; Preeclampsia Mild
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum Sample (10 mL) Plasma Sample (10 mL) Urine Collection Saliva Swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to

1. Identify a cut-off for the ratio of the serum proteins soluble FMS-like Tyrosine Kinase 1 (sFLT-1) and placental growth factor (PlGF) that identifies women will who develop preeclampsia with severe features within 2 weeks of testing (clinically positive) from those who do not develop preeclampsia with severe features within 2 weeks of testing (clinically negative) among preterm pregnant women with hypertensive disorders of pregnancy.

   And
2. To validate the cut-off the ratio of sFLT-1 and PlGF and to validate the performance of the automated assays used to find the cut-off. Test performance includes positive predictive value, negative predictive value, sensitivity, and specificity.

Subjects will provide blood, urine, and saliva samples at the time of enrollment. Samples will be frozen for batch assessment of sFLT-1 and PlGF levels by automated assays. Clinicians, subjects, and researchers will be blinded to protein level assessment, therefore assay results will not affect clinical management.

DETAILED DESCRIPTION:
Preeclampsia is a leading cause of maternal and fetal morbidity and mortality in the US, and affects about 5% of pregnancies. Despite its morbidity, preeclampsia is challenging to distinguish from worsening chronic hypertension or gestational hypertension. Furthermore, it is challenging to identify who among those with hypertensive disorders of pregnancy will develop preeclampsia with severe features, including kidney, liver, pulmonary, or cerebral injury. The only definitive treatment is delivery of the placenta, and therefore the fetus, which can lead to severe morbidity and mortality to the neonate if delivery is very premature. New methods of risk stratification are needed to identify who among women with hypertensive disorders of pregnancy are at risk of developing preeclampsia with severe features in order to allocate resources (e.g. betamethasone and magnesium for fetal neuroprotection) accordingly.

Several serum proteins (sFLT-1 and PlGF) correlate well with the development of preeclampsia, particularly with preeclampsia with severe features, and may be used to predict the development of preeclampsia with severe features within a certain timeframe. The goal of this study is to identify a cut-off of the sFLT-1/PlGF ratio using automated assays that differentiates women who will develop preeclampsia with severe features from those who will not among women with hypertensive disorders of pregnancy within 2 weeks of testing. The secondary outcomes include time to delivery, the performance of the cut-off to predict adverse maternal and adverse fetal outcomes, and a comparison of the performance of the cut-off with clinical and laboratory factors per American College of Obstetricians and Gynecologists (ACOG) guidelines. Investigators will also look at the levels of sFLT-1 and PlGF in the urine and the saliva to determine if they correlate well with serum levels and may provide a less invasive alternative to serum samples.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a pregnant woman ≥ 18 years of age.
* Gestational age 23+0 to 34+6/7 weeks
* Singleton pregnancy
* Hospitalized with (or develop while hospitalized) a hypertensive disorder of pregnancy (preeclampsia, chronic hypertension with or without superimposed preeclampsia or gestational hypertension) as defined by ACOG guidelines.

Exclusion Criteria:

* 1. Patients who have received intravenous heparin within 24 hours of enrollment. Low dose subcutaneous heparin or low molecular weight heparin (LMWH) for prophylaxis of deep venous thrombosis (DVT) is permitted.
* Patients who are currently participating in another clinical trial to evaluate a new therapeutic intervention or who have participated in another such trial in the previous 30 days.
* Multiple gestations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes women with singleton pregnancies at 23+0 to 34+6/7 weeks gestational age who are hospitalized with (or develop while hospitalized) a hypertensive disorder of pregnancy. Minors and patients who have received intravenous heparin within 24 hours of enrollment or who have participated in a therapeutic interventional study in the last 30 days will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Derivation and Performance of Cut-off for sFLT-1/PlGF Ratio (Serum) | 2 weeks
  Identification of the cut-off and performance (sensitivity, specificity, positive predictive value, and negative predictive value) for the sFLT-1/PlGF ratio as determined by automated assays that enable differentiation of those women with a hypertensive disorder of pregnancy who develop preeclampsia with severe features from those who do not develop preeclampsia within 2 weeks of testing.
Validation of Cut-off and Performance of sFLT-1/PlGF Ratio as Defined in Derivation Cohort (Serum) | 2 weeks
  Validation of the performance (sensitivity, specificity, positive predictive value, negative predictive value) of the cut-off of the sFLT-1/PlGF ratio differentiating the development of preeclampsia with severe features within 2 weeks after testing as determined by the independent Derivation cohort.

SECONDARY OUTCOMES:
Performance in Determining the Risk for Adverse Maternal Outcomes | 2 weeks
  Performance (sensitivity, specificity, positive predictive value, negative predictive value) of the sFLT-1/PlGF cut-off identified and validated per primary endpoint in determining the risk of adverse maternal outcomes within 2 weeks after testing.
Performance in Determining the Risk for Adverse Fetal/Neonatal Outcomes | 4 weeks
  Performance (sensitivity, specificity, positive predictive value, negative predictive value) of the sFLT-1/PlGF cut-off identified and validated per primary endpoint in determining the risk of adverse fetal/neonatal outcomes within 2 weeks after testing.
Performance As Compared to ACOG-Guidelines | 2 years
  Performance of the sFLT-1/PlGF ratio versus the performance of clinical and laboratory factors per ACOG guidelines in predicting maternal development of preeclampsia with severe features.
  ACOG guidelines in predicting the development of preeclampsia include,
  * systolic blood pressure of 140 mm Hg or more or diastolic blood pressure of 90 mm HG or more on at least 2 occasions at least 4 hours apart
  * 300 mg or more of protein per 24 hour urine collection
  * Protein/creatinine ration of 0.3 mg/dL or more
  * Urine dipstick reading of 2+
  * Uric acid greater than 5 mg/dL
Performance of sFLT-1/PlGF & ACOG Guidelines | 2 years
  Performance of the algorithm combining the sFLT-1/PlGF ratio PLUS clinical and laboratory factors per ACOG guidelines in predicting maternal development of preeclampsia with severe features.
  ACOG guidelines in predicting the development of preeclampsia include,
  * systolic blood pressure of 140 mm Hg or more or diastolic blood pressure of 90 mm HG or more on at least 2 occasions at least 4 hours apart
  * 300 mg or more of protein per 24 hour urine collection
  * Protein/creatinine ration of 0.3 mg/dL or more
  * Urine dipstick reading of 2+
  * Uric acid greater than 5 mg/dL
Time to Delivery | 2 years
  Time to delivery in women whose sFLT-1/PlGF ratio is above the cut-off as identified per the primary objective compared to those whose sFLT-1/PlGF ratio is below that cut-off.
sFLT-1 and PlGF Levels in Urine and Saliva | 2 years
  Identification of levels of sFLT-1 (pg/ml) and PlGF (pg/ml) in urine and saliva specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Ananth Karumanchi, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (18):
- United States (18):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - UC San Francisco Medical Center, San Francisco, California
  - Torrance Memorial Medical Center, Torrance, California
  - University of South Florida, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Northshore, Evanston, Illinois
  - MedStar Health, Baltimore, Maryland
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of North Carolina Medical Center- Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Levine RJ, Maynard SE, Qian C, Lim KH, England LJ, Yu KF, Schisterman EF, Thadhani R, Sachs BP, Epstein FH, Sibai BM, Sukhatme VP, Karumanchi SA. Circulating angiogenic factors and the risk of preeclampsia. N Engl J Med. 2004 Feb 12;350(7):672-83. doi: 10.1056/NEJMoa031884. Epub 2004 Feb 5. PMID 14764923
- [Background] Sunderji S, Gaziano E, Wothe D, Rogers LC, Sibai B, Karumanchi SA, Hodges-Savola C. Automated assays for sVEGF R1 and PlGF as an aid in the diagnosis of preterm preeclampsia: a prospective clinical study. Am J Obstet Gynecol. 2010 Jan;202(1):40.e1-7. doi: 10.1016/j.ajog.2009.07.025. Epub 2009 Sep 17. PMID 19762001
- [Background] Engels T, Pape J, Schoofs K, Henrich W, Verlohren S. Automated measurement of sFlt1, PlGF and sFlt1/PlGF ratio in differential diagnosis of hypertensive pregnancy disorders. Hypertens Pregnancy. 2013 Nov;32(4):459-73. doi: 10.3109/10641955.2013.827205. Epub 2013 Aug 19. PMID 23957293
- [Background] Verlohren S, Herraiz I, Lapaire O, Schlembach D, Moertl M, Zeisler H, Calda P, Holzgreve W, Galindo A, Engels T, Denk B, Stepan H. The sFlt-1/PlGF ratio in different types of hypertensive pregnancy disorders and its prognostic potential in preeclamptic patients. Am J Obstet Gynecol. 2012 Jan;206(1):58.e1-8. doi: 10.1016/j.ajog.2011.07.037. Epub 2011 Jul 30. PMID 22000672
- [Background] Rana S, Powe CE, Salahuddin S, Verlohren S, Perschel FH, Levine RJ, Lim KH, Wenger JB, Thadhani R, Karumanchi SA. Angiogenic factors and the risk of adverse outcomes in women with suspected preeclampsia. Circulation. 2012 Feb 21;125(7):911-9. doi: 10.1161/CIRCULATIONAHA.111.054361. Epub 2012 Jan 18. PMID 22261192
- [Background] Zeisler H, Llurba E, Chantraine F, Vatish M, Staff AC, Sennstrom M, Olovsson M, Brennecke SP, Stepan H, Allegranza D, Dilba P, Schoedl M, Hund M, Verlohren S. Predictive Value of the sFlt-1:PlGF Ratio in Women with Suspected Preeclampsia. N Engl J Med. 2016 Jan 7;374(1):13-22. doi: 10.1056/NEJMoa1414838. PMID 26735990
- [Derived] Thadhani R, Lemoine E, Rana S, Costantine MM, Calsavara VF, Boggess K, Wylie BJ, Moore Simas TA, Louis JM, Espinoza J, Gaw SL, Murtha A, Wiegand S, Gollin Y, Singh D, Silver RM, Durie DE, Panda B, Norwitz ER, Burd I, Plunkett B, Scott RK, Gaden A, Bautista M, Chang Y, Diniz MA, Karumanchi SA, Kilpatrick S. Circulating Angiogenic Factor Levels in Hypertensive Disorders of Pregnancy. NEJM Evid. 2022 Dec;1(12):EVIDoa2200161. doi: 10.1056/EVIDoa2200161. Epub 2022 Nov 9. PMID 38319832